CLINICAL TRIAL: NCT06067984
Title: A Single-Arm, Open Label, 16-week Extension Study to Evaluate the Efficacy and Safety of a Second Course of a Digital Therapeutic as an Adjunct to Standard of Care Antipsychotic Therapy in Adult and Late Adolescent Participants With Experiential Negative Symptoms of Schizophrenia
Brief Title: An Extension Study of a Second Course of a Digital Therapeutic for the Treatment of Experiential Negative Symptoms of Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-155-E-001
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Negative Symptoms in Schizophrenia
Keywords: Prescription digital therapeutic (PDT); Software as a Medical Device (SaMD); Smartphone app; Schizophrenia; Negative Symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: This study evaluates the efficacy of a prescription digital therapeutic (PDT) in addition to standard of care (SOC) therapy for the treatment of experiential negative symptoms of schizophrenia in late adolescents and adults.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Arm A (Experimental): Evaluate the efficacy and safety of a digital therapeutic as an adjunct treatment to SOC in participants with experiential negative symptoms of schizophrenia.
  Interventions: Device: Study App

INTERVENTIONS:
Device: Study App — An investigational prescription digital therapeutic in the form of a smartphone app.

SUMMARY:
The purpose of the proposed an open label extension (OLE) study is to evaluate the maintained efficacy and safety of a second consecutive course of Click Therapeutics Study App as an adjunct treatment to standard of care (SOC) in participants who were on the Study App and have recently completed the Click Therapeutics Randomized Clinical Trial NCT05838625.

DETAILED DESCRIPTION:
Click Therapeutics Study App is an interactive, software-based intervention for experiential negative symptoms of schizophrenia.

The purpose of the proposed OLE study is to evaluate the maintained efficacy and safety of a second consecutive course of Click Therapeutics Study App as an adjunct treatment to standard of care (SOC) in participants who were on the Study App and have recently completed the Click Therapeutics Randomized Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for entry into the study if all the following criteria are met:

* Completed participation in NCT05838625 study within 7 days of the extension study Baseline Visit (Day 1).
* Is the sole user of an iPhone with an iPhone operating system (iOS) 14 or greater or a smartphone with an Android operating system (OS) 10 or greater and is willing to download and use the specified Study App required by the protocol.
* Is willing and able to receive SMS text messages and push messages on their smartphone.
* It is the owner of, and has regular access to, an email address.
* Has regular access to the Internet via cellular data plan and/or wi-fi.
* Had stable housing during NCT05838625, with no anticipated housing changes during the duration of this study.

Exclusion Criteria:

A participant will not be eligible for study entry if any of the following criteria are met:

* Has not completed the Week 16 Visit (Day 112) in the NCT05838625 study.
* Has a positive urine drug screening or participant self-reports use of synthetic cathinones (bath salts), synthetic cannabinoids (K2, Spice), inhalants, amphetamines (including MDMA/ecstasy), phencyclidine (PCP), cocaine, opiates, benzodiazepines, barbiturates, hallucinogens, or parenteral drugs. Participants with a positive urine drug test and/or recreational use of THC will not be excluded from the study at the discretion of the investigator. Participants with a positive urine drug screen (UDS) or self-report who have a valid prescription for barbiturates, benzodiazepines, or opiates will not be excluded from the study at the discretion of the investigator.
* Has suicidal ideation or behavior, as assessed by the C-SSRS:

  1. Participants with a "yes" response to either Items 4 or 5 on the C-SSRS Suicidal Ideation Item during the NCT05838625 study.
  2. Participants with a "yes" response on the C-SSRS Suicidal Behavior Items within the last 6 months (26 weeks) prior to or at the Baseline Visit
* Participants who, in the opinion of the investigator, present a serious risk of suicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Change in Experiential Negative Symptoms | Baseline to Week 16
  Change from baseline to Week 16 in the Clinical Assessment Interview for Negative Symptoms, Motivation and Pleasure Scale (CAINS-MAP)

SECONDARY OUTCOMES:
Change in Experiential Negative Symptoms | Baseline to Week 8
  Change from baseline to Week 8 in the CAINS-MAP
Change in Expressive Negative Symptoms | Baseline to Weeks 8 and 16
  Change from baseline to Week 8 and to Week 16 in expressive negative symptoms, as assessed by the CAINS-EXP
Change in Positive Symptoms | Baseline to Week 16
  Change from baseline to Week 16 in positive symptoms, as assessed by the Positive and Negative Syndrome Scale (PANSS)
Change in Social Functioning | Baseline to Week 16
  Change from baseline to Week 16 in social functioning, as assessed by the Personal and Social Performance Scale (PSP)
Change in Defeatist Beliefs | Baseline to Week 16
  Change from baseline to Week 16 in self-reported defeatist beliefs, as assessed by the Defeatist Beliefs Subscale of the Dysfunctional Attitude Scale (DAS)
Impression of Improvement | Week 16
  Patient Global Impression of Improvement Scale (PGI-I) at Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Viveca Livezey, MD, Study Director — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No